CLINICAL TRIAL: NCT02993042
Title: Effect of Robot-assisted Gait Training on Gait Automaticity in Patients With Parkinson's Disease: a Feasibility Study
Brief Title: Effect of Robot-assisted Gait Training on Gait Automaticity in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Han Gil Seo, Clinical Assistant Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAGT-GAP
Record Dates: First submitted 2016-12-06; First posted 2016-12-14 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Parkinson Disease; Gait Disorders, Neurologic
Keywords: Rehabilitation; Robot-assisted gait training
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic

ARMS (1):
- Robot-assisted gait training (Experimental): Robot-assisted gait training using an exoskeletal robot (Walkbot_S; P&S Mechanics Co. Ltd., Seoul, Korea)
  Interventions: Device: Robot-assisted gait training

INTERVENTIONS:
Device: Robot-assisted gait training — Patients should use their belts (Harness) to support their weight when walking in equipment. In the first training session, the patient focuses on fitting and adapting the equipment and helps the patient learn. To minimize skin damage, the patient can wear a protector. The initial walking speed starts at 1.5km / h (0.42m / s) and can be increased gradually to 3.0km / h (0.83m / s) by increasing to 0.2km / h (0.06m / s) per session. The therapist provides appropriate visual and auditory instructions to allow the patient to participate as fully as possible in the walking cycle provided by the walking robot. The treatment time per session is 30 minutes except for the time of wearing and releasing.

SUMMARY:
Robot-assisted gait training can improve gait ability of patients with Parkinson's disease by repeating a normal gait pattern with high intensity. This study is a feasibility study to investigate whether robot-assisted gait training can be applied to improve walking autonomy in patients with Parkinson 's disease.

DETAILED DESCRIPTION:
Parkinson's disease is a disease caused by dopamine deficiency in the striatum resulting from the loss of dopaminergic neuronal cells in the cerebral substantia. It is a progressive neurodegenerative disease characterized by motor symptoms including gait disturbance and balance instability. In the early stages of Parkinson's disease, dysfunction of the sensorimotor area of the basal ganglia typically occurs, leading to habitual control hurdles. Accordingly, cognitive efforts are required to perform habitual tasks such as walking, and the automaticity of walking is reduced. Walking performance in a dual-task condition has been used to assess gait automaticity in patients with Parkinson's disease.

Robot-assisted gait training is a method of rehabilitation that repeats normal gait patterns at high intensity. Recent meta-analysis has shown that robot-assisted gait training improved the recovery of independent gait after stroke compared with conventional rehabilitation therapy. On the other hand, robot-assisted gait training in Parkinson's disease has been reported to improve walking speed and walking endurance compared to conventional physical therapy, but is not superior to treadmill exercise of the same intensity. In addition, it has been reported that in patients with Parkinson's disease with balance impairment, robot-assisted gait training can improve balance disorder compared with physical therapy, and gait freezing has improved in some small-scale patients. However, studies on the effectiveness of robot-assisted gait training in Parkinson's disease are still lacking, and the mechanism of the effect has not been elucidated. In particular, the effect on gait automaticity, which is a characteristic of Parkinson 's disease, has not been studied. Therefore, this pilot study is aimed to investigate whether robot-assisted gait training can be applied to improve walking autonomy in patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed patients with idiopathic Parkinson's disease
* Hoehn & Yahr stage 2.5 or 3 patients
* Patients with a Mini-Mental Status Examination (MMSE) score of 24 or higher

Exclusion Criteria:

* Patients with severe dyskinesia or on-off fluctuations due to medication
* Patients who need to change drugs during the study period
* Patients with sensory abnormalities of the lower limb
* Patients with vestibular disease or paroxismal vertigo
* Patients with other neurological or orthopedic disease involving legs, or severe cardiovascular diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-12; Primary Completion 2018-01 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Percentage of dual-task interference: cognitive | at 4 weeks
  (Cognitive dual-task performance - Single-task performance) / Single-task performance during 10 meter walk test
Percentage of dual-task interference: physical | at 4 weeks
  (Physical dual-task performance - Single-task performance) / Single-task performance during 10 meter walk test

SECONDARY OUTCOMES:
10 meter walk test (sec): single, cognitive dual-task, physical dual-task | baseline, at 4 weeks, at 8 weeks
Berg balance scale | baseline, at 4 weeks, at 8 weeks
Korean version of the Falls Efficacy Scale-International | baseline, at 4 weeks, at 8 weeks
Step length | baseline, at 4 weeks, at 8 weeks
  Gait analysis using IMU sensors
Step width | baseline, at 4 weeks, at 8 weeks
  Gait analysis using IMU sensors
Cadence | baseline, at 4 weeks, at 8 weeks
  Gait analysis using IMU sensors
Vertical displacement | baseline, at 4 weeks, at 8 weeks
  Gait analysis using IMU sensors
Percentage of dual-task interference: cognitive | baseline, at 8 weeks
  (Cognitive dual-task performance - Single-task performance) / Single-task performance during 10 meter walk test
Percentage of dual-task interference: physical | baseline, at 8 weeks
  (Physical dual-task performance - Single-task performance) / Single-task performance during 10 meter walk test

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea